CLINICAL TRIAL: NCT06278402
Title: Efficacy of Oral Tofacitinib in Moderate to Severe Alopecia Areata, Totalis and Universalis at Tertiary Care Hospital, Karachi.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jinnah Hospital (Other)
Responsible Party: Principal Investigator, Misbah Zari Qadir, Principal Investigator, Jinnah Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JinnahH
Record Dates: First submitted 2024-01-28; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Alopecia Areata; Alopecia Totalis; Alopecia Universalis
Keywords: Tofacitinib; Alopecia areata; Janus kinase inhibitor; JAK 1/3 inhibitor
MeSH Terms: conditions — Alopecia Areata; Alopecia universalis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: This study includes patients with moderate to severe Alopecia Areata, totalis and universalis. The efficacy of JAK 1/3 inhibitor, Tofacitinib will be assessed by using SALT score (Severity of Alopecia Tool) at Baseline, 06 weeks, 12 weeks and 24 weeks. Oral Tofacitinib given at a dose of 5 mg twice daily after relevant investigations. The data will be analyzed in SPSS version 23.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tofacitinib (Experimental): tofacitinib 5mg twice daily for 6 months
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Oral tofacitinib 5mg twice daily for treatment of alopecia areata, totalis and universalis.

SUMMARY:
To determine the efficacy of oral Tofacitinib in the treatment of moderate to severe alopecia areata, totalis and universalis at tertiary care hospital of Karachi, Pakistan. Efficacy of treatment in patients presenting with alopecia areata will be assessed using SALT Score on follow up at 6,12 and 24 weeks where four categories of treatment response were defined: 0 (re-growth ≤10%), 1 (11-25%), 2 (26-50%), 3 (51-75%) and 4 (re-growth >75%). Efficacy will be considered if re-growth ≥ 2.

DETAILED DESCRIPTION:
Alopecia areata is a chronic, autoimmune, non-scarring alopecia that involves the destruction of hair follicles (HF) by autoreactive CD8+ T cells. AA can affect any hair-bearing region and can manifest in various patterns ranging from patchy diffuse alopecia to progression to more severe forms such as alopecia totalis (AT) or alopecia universalis (AU). As a common type of alopecia in human, the estimated prevalence of AA is approximately between 0.1% and 0.2%, second only to male and female pattern alopecia. Although it is not life threatening but the psychosocial impact of the disease is a concern. The treatment of advanced forms of alopecia areata (AA) is more challenging than the milder forms and patients with advanced AA often require systemic therapy in order to regrow hair.

Current treatments include steroids (intralesional, topical, and systemic), topical immunotherapy (diphenylcyclopropenone [DPCP], squaric acid dibutylester [SADBE]), topical immunosuppressants (tacrolimus, pimecrolimus), topical minoxidil, and topical prostaglandin analogs (bimatoprost, latanoprost).

Significant breakthroughs in understanding of intracellular cytokine signaling pathways have promoted a dawn of new promising therapeutic agents, known as Janus kinase inhibitors (JAKs), which block signaling of certain cytokines by inhibiting ATP binding within the phosphorylation sites of cytokine receptor homo- or heterodimers, thereby interrupting the JAK/signal transducer and activator of transcription (STAT) pathway and subsequently production of pro-inflammatory cytokines and other mediators associated with AA.

Despite the rapid development of novel JAK inhibitors, including baricitinib and ritlecitinib, tofacitinib remains an effective and the longest-used JAK inhibitor for AA. Tofacitinib primarily targets JAK 1/3 and reduces the immune response and resultant inflammation, emerging as an alternative for the treatment of refractory cases of AA.

In 2014, the first reported case using a JAK1/3 inhibitor, tofacitinib citrate, for the treatment of AU was described in a patient with concomitant plaque psoriasis who achieved full regrowth of hair within 8 months. Since then, the scientific understanding of AA has continued to progress, highlighting the key role that cytotoxic T lymphocytes play in AA and the potential of JAK inhibition. Due to the lack of data regarding efficacy and safety of this drug in alopecia areata we therefore aim to provide a comprehensive literature, evaluate the effectiveness, outcome and role of Tofacitinib in the treatment of AA.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with Alopecia areata as per operational definition will be included in the study.
* Either gender.
* Age 15 - 60 years.

Exclusion Criteria:

* Patient with history of connective tissue disorders, vasculitis, seropositive and seronegative arthritis.
* Patients having history of treatment with systemic agents, having active infection, pregnant and lactating women and patients having severe hematological abnormalities.
* Patients positive for latent infections.
* Patients with weight <25 kg.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-01-06 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Alopecia | 6 months
  To analyze the efficacy of oral Tofacitinib in moderate to severe alopecia areata, totalis and universalis at Tertiary Care Hospital, Karachi. The effect of treatment will be evaluated using photographs of the patient before and after the trial and clinical evaluation of patients. The clinical response for efficacy will be evaluated at 0, 6,12 and 24 weeks of therapy. Patient presenting with alopecia areata will be assessed for degree of improvement using SALT score on follow up after 3 months as follows: 0 (re-growth ≤10), 1 (11-25%), 2 (26-50%), 3 (51-75%) and 4 (re-growth >75%). Efficacy will be considered if re-growth ≥3.

CONTACTS AND LOCATIONS:
Locations (1):
- Misbah Zari Qadir, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Literature review, statistical analysis of efficacy of tofacitinib in the treatment of alopecia areata, totalis and universalis.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Result] Husein-ElAhmed H, Abdulla N, Al-Obaidli A, Ali-Alam M, Steinhoff M. Real-world experience and long-term evaluation of tofacitinib in refractory alopecia areata: A prospective, open-label, single-center study in Asian Arab population. Dermatol Ther. 2022 Dec;35(12):e15871. doi: 10.1111/dth.15871. Epub 2022 Dec 1. PMID 36177791
- [Result] Sardana K, Bathula S, Khurana A. Which is the Ideal JAK Inhibitor for Alopecia Areata - Baricitinib, Tofacitinib, Ritlecitinib or Ifidancitinib - Revisiting the Immunomechanisms of the JAK Pathway. Indian Dermatol Online J. 2023 Jun 28;14(4):465-474. doi: 10.4103/idoj.idoj_452_22. eCollection 2023 Jul-Aug. PMID 37521227
- [Result] Dillon KL. A Comprehensive Literature Review of JAK Inhibitors in Treatment of Alopecia Areata. Clin Cosmet Investig Dermatol. 2021 Jun 25;14:691-714. doi: 10.2147/CCID.S309215. eCollection 2021. PMID 34211288
- [Result] Pratt CH, King LE Jr, Messenger AG, Christiano AM, Sundberg JP. Alopecia areata. Nat Rev Dis Primers. 2017 Mar 16;3:17011. doi: 10.1038/nrdp.2017.11. PMID 28300084
- [Result] Donovan J. The Evolving Story of JAK Inhibitors for Treating Alopecia Areata: A Review of Current Progress and Future Directions. Skin Therapy Lett. 2023 May;28(3):1-7. PMID 37339501
- [Result] Gupta AK, Carviel JL, Foley KA, Shear NH, Piraccini BM, Piguet V, Tosti A. Monotherapy for Alopecia Areata: A Systematic Review and Network Meta-Analysis. Skin Appendage Disord. 2019 Nov;5(6):331-337. doi: 10.1159/000501940. Epub 2019 Aug 29. PMID 31799258
- [Result] Huang J, Deng S, Li J, Tang Y, Liu F, Liu Y, Rao S, Shi W. Drug Survival and Long-term Outcome of Tofacitinib in Patients with Alopecia Areata: A Retrospective Study. Acta Derm Venereol. 2023 Nov 13;103:adv13475. doi: 10.2340/actadv.v103.13475. PMID 37955531
- [Result] Damsky W, King BA. JAK inhibitors in dermatology: The promise of a new drug class. J Am Acad Dermatol. 2017 Apr;76(4):736-744. doi: 10.1016/j.jaad.2016.12.005. Epub 2017 Jan 28. PMID 28139263
- [Result] Craiglow BG, King BA. Killing two birds with one stone: oral tofacitinib reverses alopecia universalis in a patient with plaque psoriasis. J Invest Dermatol. 2014 Dec;134(12):2988-2990. doi: 10.1038/jid.2014.260. Epub 2014 Jun 18. No abstract available. PMID 24940651
- [Result] Liu LY, King BA. Tofacitinib for the Treatment of Severe Alopecia Areata in Adults and Adolescents. J Investig Dermatol Symp Proc. 2018 Jan;19(1):S18-S20. doi: 10.1016/j.jisp.2017.10.003. PMID 29273099